CLINICAL TRIAL: NCT02162147
Title: How Safe Are Our Pediatric Emergency Departments? A National Prospective Cohort Study
Brief Title: How Safe Are Our Pediatric Emergency Departments?
Status: Completed | Type: Observational
Sponsor: Children's Hospital of Eastern Ontario (Other)
Collaborators: Provincial Health Services Authority British Columbia (Other); Stollery Children's Hospital (Other); Alberta Children's Hospital (Other); The Children's Hospital of Winnipeg (Other); London Health Sciences Centre (Other); The Hospital for Sick Children (Other); St. Justine's Hospital (Other); Janeway Children's Health and Rehabilitation Centre (Unknown); Manitoba Institute of Child Health (Industry); Ottawa Hospital Research Institute (Other)
Responsible Party: Principal Investigator, Amy Plint, Senior Scientist, CHEO Research Institute; Physician, Division of Emergency Medicine, Children's Hospital of Eastern Ontario
Other Study IDs: 14/70X; 312463 (Other Grant/Funding Number: CIHR)
Record Dates: First submitted 2014-06-10; First posted 2014-06-12 (Estimated); Last update posted 2018-01-17 (Actual); Status verified 2018-01

CONDITIONS: Adverse Effects; Adverse Drug Event
Keywords: patient safety; pediatrics; emergency medicine
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Patient safety is an internationally recognized health care priority. Canadian data suggests that about 8% of adults admitted to hospital experience unintended harm (or 'adverse events') from the health care provided during their hospital stay. On a national level, this represents almost 25,000 preventable deaths among hospitalized adults each year. The emergency department is recognized as a high-risk environment for adverse events but most patient safety research is not specific to the emergency department. As well, the vast majority of people treated in the emergency department are sent home after their visit; yet safety research focuses primarily on people who are admitted to hospital. Finally, although children have also been identified as particularly high risk for suffering adverse events, very little research has been done on how often these events occur among children who visit the emergency department. Our study will address this gap in our knowledge about patient safety and provide important information on the frequency, severity and preventability of adverse events occurring among children in the emergency department. This information will help us to improve the safety of emergency department care for all Canadian children.

ELIGIBILITY:
Inclusion Criteria:

* Age less than 18 years
* Patients from all pediatric Canadian Triage Acuity Scale categories (pedsCTAS; 1:resuscitation; 2:emergent, 3:urgent, 4:semi-urgent, 5:non-urgent).

Exclusion Criteria:

* Insurmountable language barrier that prevents informed consent and follow-up by telephone.
* Children and families that will be unavailable for telephone follow-up in the three weeks after their emergency department visit (e.g., no telephone in the home, travelling out of the country, etc.).

Ages: 1 Day to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Subjects presenting to one the nine participating Canadian pediatric hospitals (BC Children's Hospital (BC), CHU Sainte-Justine (PQ), Children's Hospital of Eastern Ontario (ON), The Hospital for Sick Children (ON), Children's Hospital of Western Ontario (ON), Children's Hospital of Winnipeg (MB), Janeway Children's Health and Rehabilitation Centre (NL), Stollery Children's Hospital (AB) and Alberta Children's Hospital (AB)) Emergency Departments
Sampling Method: Non-Probability Sample
Enrollment: 6385 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who experience an adverse event related to emergency department care within 3 weeks of an emergency department visit | 3 weeks
  An adverse event will be defined as an event that results in unintended harm to the patient, and is related to the health care and/or services provided to the patient rather than to the patient's underlying medical condition. Emergency department care will be defined as any care provided in the emergency department and will explicitly include care provided by emergency department specific staff (i.e., staff physicians, nurses, and allied health care providers) and care provided by consultants in the emergency department.

SECONDARY OUTCOMES:
Proportion of patients experiencing a preventable adverse event | 3 weeks
Clinical severity of adverse events | 3 weeks
  For all patients, we will report the clinical severity as: (a) an abnormality on laboratory testing, (b) ≤1 day of symptoms, (c) >1 day of symptoms, (d) nonpermanent disability (e) permanent disability, or (f) death. For admitted patients, we will also report clinical severity according to The Institute for Health Care Improvement trigger tool categories: (a) temporary harm to the patient requiring intervention, (b) temporary harm to the patient requiring initial or prolonged hospitalization, (c) permanent patient harm, (d) intervention required to sustain life, or (e) death.
Types of adverse events | 3 weeks
  Adverse Events will be classified as (a) diagnostic issue, (b) management issue, (c) unsafe disposition decision, (d) suboptimal follow-up, (e) medication adverse effect, (f) procedural complication, and (g) nosocomial infection
System response required for adverse events | 3 weeks
  The response will be classified as: (a) no treatment (symptoms only), (b) required medical/surgical intervention, (c) visit to MD office, (d) Emergency Department visit, (e) admission to hospital. These previously published broad categories were chosen in order to address the effect of the Adverse Events at both the patient and health care system level.These categories are not exclusive.
Proportion of patients for whom an adverse event is related to emergency department specific care | 3 weeks
  Versus consulting specialty service care provided in the emergency department or care provided after the child's emergency department visit
Adverse events related to care provided in the emergency department by consulting service | 3 weeks
Patient and system level characteristics associated with adverse events and preventable adverse events | 3 weeks
Adverse events that occur within the 3-week time frame but are not related to care received in the emergency department | 3 weeks
  Including those related to in-hospital care and primary care

CONTACTS AND LOCATIONS:
Overall Officials: Amy Plint, MD, MSc, Principal Investigator — Children's Hospital of Eastern Ontario; Lisa Calder, MD, Principal Investigator — Ottawa Hospital Research Institute
Locations (10):
- Canada (10):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - BC Children's Hospital, Vancouver, British Columbia
  - Manitoba Institute of Child Health, Winnipeg, Manitoba
  - Winnipeg Children's Hospital, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - Children's Hospital at London Health Sciences Centre, London, Ontario
  - Children's Hospital for Eastern Ontario, Ottawa, Ontario
  - The Hospital for Sick Children, Toronto, Ontario
  - CHU Sainte-Justine, Montreal, Quebec

REFERENCES:
- [Derived] Plint AC, Newton A, Stang A, Bhatt M, Barrowman N, Calder L; Pediatric Emergency Research Canada (PERC). How safe are our paediatric emergency departments? Protocol for a national prospective cohort study. BMJ Open. 2014 Dec 4;4(12):e007064. doi: 10.1136/bmjopen-2014-007064. PMID 25475246